CLINICAL TRIAL: NCT02941575
Title: Esthetic Patient Satisfaction and Peri-Implant Tissue Success of Crystal Ultra Hybrid Ceramic Compared to E-Max Superstructures in Esthetic Zone
Brief Title: Patient Satisfaction and Peri-Implant Tissue Success of Hybrid Ceramic Versus E-Max Superstructures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Samir Bushra, Lecturer Assistance, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-215
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Implant superstructure crown: All ceramic, IPS Emax
  Interventions: Other: All ceramic
- Intervention (Experimental): Implant superstructure crown: Hybrid ceramic, crystal Ultra crown
  Interventions: Other: Crystal Ultra

INTERVENTIONS:
Other: Crystal Ultra — Crystal Ultra: is a resin nano-ceramic material, that combines both advantages of ceramics and composites.
  Other Names: hybrid ceramics, resin nanoceramic e.g Cerasmart
  Arms: Intervention
Other: All ceramic — IPS Emax: is an all ceramic crown that has proven superior aesthetics and strength properties.
  Other Names: IPS-Emax, all ceramic crowns
  Arms: Control

SUMMARY:
In patients receiving implants in the esthetic zone, would the use of new Nano hybrid ceramic crown material (Crystal Ultra) improve esthetic patient satisfaction and peri-implant tissue success when compared with Lithium Disilicate crown (E-max)?

DETAILED DESCRIPTION:
The patient will be treated in visits designated as follows:

Visit 1: Preoperative records, face-to-face adherence reminder session, signing consents, clinical, radiographic examination and primary impression for diagnostic cast construction.

Visit 2: (first stage surgery): implant placement surgical procedure and postoperative radiograph.

Visit 3: After 3months (second stage surgery): re-opening of surgical site, placement of healing abutments and temporary crowns.

Visit 4: After 2 weeks, removing of temporary restorations and taking of final impressions Visit 5: placement of different ceramic crown superstructures and recording different outcome values.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years with at least one tooth missing in the esthetic area.
2. Available bone for implant placement:

   A. Labial and Palatal Plate of bone not less than 2mm. B. Mesio- distal dimension not less than 6.5mm. C. Bone length not less than 9mm.
3. Patient with good oral hygiene.
4. Class 1 occlusion.
5. Lack of excessive parafunctional activity leading to implant failure.
6. Tooth extracted not less than 6 month.

Exclusion Criteria:

1. Young patients in whom the jaws are still growing. (Less than 18 years).
2. Jaw pathology.
3. Smokers.
4. Uncontrolled Diabetic or particularly insulin-dependent.
5. Radiotherapy to the neck or face.
6. Multiple loss of teeth which may be indicated for more complicated procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Esthetic Patient satisfaction | 1 year
  Measurement unit is Binary

SECONDARY OUTCOMES:
Peri-implant tissue success (A-Marginal Bone Loss, B-Relative attachment level, C-Peri-Implant Probing depth, D-Sulcus bleeding) | 1 year
  Measurement unit is Categorical

CONTACTS AND LOCATIONS:
Overall Officials: Jylian El Guindy, Professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No